CLINICAL TRIAL: NCT04610853
Title: Rotational Thromboelastometry Versus The Disseminated Intravascular Coagulation Score in Sepsis (RODSS)
Brief Title: Rotational Thromboelastometry Versus DIC Score in Sepsis
Acronym: RODSS
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Sirak Petros, MD, Professor, University of Leipzig
Other Study IDs: RODSS-2020
Record Dates: First submitted 2020-10-18; First posted 2020-11-02 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Sepsis; Septic Shock
Keywords: sepsis; septic shock; disseminated intravascular coagulation; rotational thromboelastometry; DIC score
MeSH Terms: conditions — Sepsis; Shock, Septic; Disseminated Intravascular Coagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Citrate plasma as a backup for coagulation profile
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: rotational thromboelastometry — ROTEM will be conducted and DIC score calculated within 24 hours after the diagnosis of Sepsis as well as on day 3 and 5 of ICU stay

SUMMARY:
Sepsis results in activation of the coagulation system, which is commonly described as disseminated intravascular coagulation (DIC). The DIC score, which is commonly used to define this syndrome, does not allow to delineate between hypercoagulation and hypocoagulation. The aim of this prospective observational study is to evaluate data from automated rotational thromboelastometry and compare These with the DIC score regarding intensive care unit outcome.

DETAILED DESCRIPTION:
Sepsis results in an intensive interaction between Inflammation and the coagulation system. The activation of the coagulation system leads to consumption of procoagulatory as well as anticoagulatory proteins and platelets. This process may induce microcirculatory thrombosis as well as hemorrhagic diathesis, which is commonly described as disseminated intravascular coagulation (DIC).

The International Society on Thrombosis and Haemostasis (ISTH) recommends the use of the DIC score to describe this syndrome. A score of at least 5 points is defined as an overt DIC. However, the DIC score does not allow to differentiate between a hypercoagulation and hypocoagulation states and whether there could be a difference regarding outcome between the two states.

In this prospective observational study, patients admitted to a medical intensive care unit will be included. The DIC score as well as rotational thromboelastometry (ROTEM) will be evaluated within the first 24 hours after the diagnosis of sepsis as well as on day 3 and 5.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis, defined according to the Sepsis-3 Definition
* informed consent

Exclusion Criteria:

* age <18 years
* pregnancy and lactation
* known coagulation disorder prior to Admission for sepsis
* known cirrhosis of the liver
* known active malignancy
* surgical procedure during the last 4 weeks
* refusal to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with sepsis admitted to a medical intensive care unit
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Correlation between the clotting time, clot formation time, maximum clot firmness and lysis index at 30 minutes from FIBTEM, INTEM, EXTEM and APTEM measurements of the ROTEM assay with an overt DIC on the day of sepsis diagnosis regarding ICU survival | through study completion, up to an average of 7 days
  The ICU survival of patients with abnormal clotting time, clot formation time, maximum clot firmness or lysis index at 30 minutes from FIBTEM, INTEM, EXTEM and APTEM of the ROTEM assay will be compared to that of patients with an overt DIC according to the criteria of the International Society on Thrombosis and Haemostasis (ISTH)

SECONDARY OUTCOMES:
correlation between ROTEM variables and the Sequential Organ Function Assessment Score | through study completion, up to an average of 7 days
  The Sequential Organ Function Assessment (SOFA) score of patients with any abnormal ROTEM variable will be compared to the score of patients without any abnormal ROTEM variable

CONTACTS AND LOCATIONS:
Overall Officials: Sirak Petros, MD, Principal Investigator — University of Leipzig
Locations (1):
- University Hospital of Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided